CLINICAL TRIAL: NCT05276414
Title: Circulating Cathodic Antigen Test Compared to Microscopy for Diagnosis of Urinary Schistosomiasis in Sohag
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Kamal Abdellah, lecturer of medical parasitology, faculty of medicine, Sohag University
Other Study IDs: Soh-Med-22-02-31
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Urinary Schistosomiases
MeSH Terms: conditions — Schistosomiasis haematobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Schistosomiasis is a chronic infection endemic in 74 tropical and sub-tropical countries. Sub-Saharan Africa carries the highest burden (90%) of schistosomiasis which caused by both Schistosoma mansoni and Schistosoma haematobium. The prevalence of Schistosomiasis should be assessed to control of the infection. This is usually achieved through surveys based on the use of traditional parasitological methods as urine filtration for S. haematobium. However, these traditional methods are time consuming, require an experienced technician and multiple samples due to light-infection and irregular shedding. Therefore, the point-of-care Circulating Cathodic Antigen (POC-CCA) urine test has been developed for the diagnosis of S. haematobium infection which is simple, rapid, sensitive and specific assay.

ELIGIBILITY:
Inclusion Criteria:

* 100 outpatient children aged between 5 - 16 years

Exclusion Criteria:

* Outpatient children should not have received schistosomiasis treatment (within the past 6 months) prior to the study

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Samples will be collected from outpatient children aged between 5 - 16 years from Pediatric outpatient Clinics in Sohag hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
to evaluate the accuracy of rapid immunochromatographic assay (POC-CCA) compared with traditional microscopic examination for diagnosis of Schistosoma haematobium infection | 16 weeks following the startpoint of the study.
  comparing the sensitivity and specificity of rapid immunochromatographic assay with traditional microscopic examination for diagnosis of Schistosoma haematobium infection

SECONDARY OUTCOMES:
to estimate the prevalence of Schistosoma haematobium infection in outpatient children in Sohag | 16 weeks following the startpoint of the study.
  By examining the stool samples of 100 outpatient children and recording the number of cases with Schistosoma haematobium infection.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa K Abd Ellah, lecturer, Principal Investigator — Medical Parasitology, Faculty of Medicine, Sohag University
Locations (1):
- Faculty of medicine,Sohag University, Sohag, Egypt